CLINICAL TRIAL: NCT01994434
Title: Ulnar Nerve Deep Branch Compression by a Ganglion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TSWang9804; HEBEI-J0821 (Other: Hebei Ethics Committee)
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2012-08

CONDITIONS: Guyon's Canal; Nerve Compression
Keywords: Deep branch of the ulnar nerve; Distal ulnar nerve compression
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decompression of the ulnar nerve (Other): Surgical decompression of the Guyon's canal and ganglion excision
  Interventions: Procedure: Decompression of the ulnar nerve

INTERVENTIONS:
Procedure: Decompression of the ulnar nerve — Surgical decompression of the Guyon's canal and ganglion excision

SUMMARY:
Ulnar nerve compression is common at the elbow, but less common at the wrist. The purposes of this study are to report a series of 9 patients with pure ulnar nerve deep branch compression by a ganglion and to evaluate the outcome following a surgical treatment. According modified Bishop's scoring system, the investigators would evaluate postoperative results of this uncommon nerve lesion.

DETAILED DESCRIPTION:
Pre- and post-operative physical examination include assessment of tenderness and strength (grip and pinch). Grip strength and tip pinch strength between the thumb and index finger are measured using the E-LINK system. According Bishop's scoring system, the investigators redesign a questionnaire for comprehensive assessment of this uncommon nerve lesion.

ELIGIBILITY:
Inclusion Criteria:

Ulnar nerve deep branch compression by a ganglion -

Exclusion Criteria:

Ulnar nerve deep branch compression caused by other reasons

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2000-03; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Grip strength | 18-24 months
  Grip strength is measured using the E-LINK system.
Tip pinch strength | 18-24 months
  Tip pinch strength between the thumb and index finger is measured using the E-LINK system.

SECONDARY OUTCOMES:
Modified Bishop's scoring system | 18-24 months
  According Bishop's scoring system, we redesign a questionnaire for comprehensive assessment of this uncommon nerve lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Almeida V, de Carvalho M. Lesion of the deep palmar branch of the ulnar nerve: causes and clinical outcome. Neurophysiol Clin. 2010 Jun;40(3):159-64. doi: 10.1016/j.neucli.2010.01.005. Epub 2010 Feb 17. PMID 20513615